CLINICAL TRIAL: NCT06092021
Title: Obesity Phenotypes and Its Relation to Cardiovascular Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Khaled Sayed, Asmaa khaled sayed, Assiut University
Other Study IDs: Cardiovascular obesity
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Cardiovascular Diseases
Keywords: Cardiovascular diseases; Obesity phenotypes
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the association between obesity phenotypes with cardiovascular diseases.

* Primary Outcomes:

  1- To examine the association between different obesity phenotypes and cardiovascular diseases.by using echocardiography, lipid profile
* Secondary Outcomes:

  1. frequency of obesity phenotypes on our locality
  2. Correlation between each type of obesity phenotypes and other metabolic disturbances (e.g. DM, dyslipidemia, NASH)
  3. Correlation between epcardial fat, carotid intimal thickness and different obesity phenotypes.

DETAILED DESCRIPTION:
Obesity is a condition caused by increasing the fat components of body resulting in body weight increase. Obesity leads to several complications like type 2 diabetes, hypertension and cardiovascular events, sleep apnea. But obesity can no longer be evaluated solely by the body mass index (expressed in kg/m2) because it represents a heterogeneous entity (1). As there are several cardio-metabolic imaging studies have shown that some individuals who have a normal weight or who are overweight are at high risk if they have an excess of visceral adipose tissue-a condition often accompanied by accumulation of fat in normally lean tissues (ectopic fat deposition in liver, heart, skeletal muscle, etc.) (2) On the other hand, individuals who are overweight or obese can nevertheless be at much lower risk than expected when faced with excess energy intake if they have the ability to expand their subcutaneous adipose tissue mass, particularly in the gluteal-femoral area, as preferential fat storage in the lower body depot may act as a metabolic buffer and protect other tissues from lipotoxicity caused by lipid overflow and ectopic fat (3). Hence, excessive amounts of visceral adipose tissue and of ectopic fat largely define the cardiovascular disease risk of overweight and moderate obesity (4). Epicardial fat is considered as indicator of cardiovascular risk. Several studies have tested the association between epicardial fat thickness (EFT) and coronary artery disease many studies stated that epicardial fat is independently and linearly associated with CAD and its severity .In this study we aim to monitor the extent of obesity phenotypes association to cardiovascular diseases in patients attending to Obesity Clinic in Assuit Hospital University.

ELIGIBILITY:
Inclusion Criteria:

- Adult patient of 18 years old and above

Exclusion Criteria:

* 1- Patients below 18 years old age (pediatrics and Child).

  2- Pregnant females.

  3- Patients with congenital heart diseases.

  4- Patients with previous bariatric surgery.

  5-Patients with type 1 DM.

  6-Patients with hereditary hyperlipidemia

  .Secondary causes of obesity

include these:Endocrine DisordersCushing SyndromeHypothyroidismPseudohypoparathyroidismType 2 diabetes

Genetic SyndromesPrader-Willi syndromeBardet-Biedel syndromeCohen syndromeCentral Nervous System DisordersHypothalamic TumorTrauma to or inflammation of the hypothalamic regionOtherDrug induced - atypical anti-psychotics, tricyclic antidepressantsBinge eating disorderBulimia nervosa

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Different obesity phenotypes people Accor to body mass index, waist circumference, waist hip ratio ,and metabolic profiles
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To examine the association between different obesity phenotypes and cardiovascular by using lipid profile and echocardiography | One year
  Using echocardiography and lipid profile to determine the relationship between obesity and cardiovascular diseases in obese and non obese people
Assess carotid artery elasticity in obese by using echocardiography | One year
  Find out the effect of cardiovascular diseases and obesity on carotid artery elasticity and atherosclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Sayed, Resident, Principal Investigator — Assiut University
Locations (1):
- Asmaa khaled sayed, Asyut, Egypt

REFERENCES:
- [Background] Vecchie A, Dallegri F, Carbone F, Bonaventura A, Liberale L, Portincasa P, Fruhbeck G, Montecucco F. Obesity phenotypes and their paradoxical association with cardiovascular diseases. Eur J Intern Med. 2018 Feb;48:6-17. doi: 10.1016/j.ejim.2017.10.020. PMID 29100895
- [Background] Piche ME, Tchernof A, Despres JP. Obesity Phenotypes, Diabetes, and Cardiovascular Diseases. Circ Res. 2020 May 22;126(11):1477-1500. doi: 10.1161/CIRCRESAHA.120.316101. Epub 2020 May 21. PMID 32437302